CLINICAL TRIAL: NCT06490796
Title: Which Respiratory Training is More Effective in Individuals with Ankylosing Spondylitis: 360-Degree Expandable Diaphragm Exercises or Standard Diaphragm Exercises? a Randomized Controlled Trial
Brief Title: Respiratory Training in Individuals with Ankylosing Spondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir University of Economics (Other)
Responsible Party: Principal Investigator, Seda Yakit Yesilyurt, Assist Prof., Izmir University of Economics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: B.30.2.İEÜSB.0.05.05-20-279
Record Dates: First submitted 2024-06-07; First posted 2024-07-08 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-07

CONDITIONS: Ankylosing Spondylitis; Exercise Training; Diaphragm; Mobility
Keywords: Ankylosing Spondylitis; Breathing; Mobility; Functional capacity; Physiotherapy
MeSH Terms: conditions — Spondylitis, Ankylosing; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Expanded diaphragm exercise arm (Experimental): participants will use Ohmbelt device during 360-degree expansive diaphragm exercise session.
  Interventions: Behavioral: Expanded diaphragm exercise
- Standard diaphragm exercise arm (Active Comparator): participants will attend standard breathing exercise sessions.
  Interventions: Behavioral: Standard diaphragm exercise

INTERVENTIONS:
Behavioral: Expanded diaphragm exercise — Individuals will be instructed in 360-degree expansive diaphragm exercises using the Ohmbelt device (Nilus Medical LLC, OHMBELT, Redwood City, CA, USA). Two Ohmbelt devices will be used in this study. The placement of the devices will be as described in the literature (14,23,24): The patient will be in a seated position with hips and knees flexed at 90 degrees, both feet supported on the ground, and sitting upright on a chair without back support. In this position, the Ohmbelt devices will be secured to the patient's body. Following respiratory exercises, they will be individually enrolled in the evidence-based consensus program for three-dimensional functional exercises recommended for AS patients (26,27). The exercise protocol, which includes warm-up, mobility, stretching, flexibility, and cool-down periods, will last for 20 minutes
  Arms: Expanded diaphragm exercise arm
Behavioral: Standard diaphragm exercise — Individuals in this group will be instructed in standard diaphragm exercises. They will be asked to lie on their backs with their heads and knees supported by pillows, and to close their eyes to focus before starting. Following respiratory exercises, they will be individually enrolled in the evidence-based consensus program for three-dimensional functional exercises recommended for AS patients (26,27). The exercise protocol, which includes warm-up, mobility, stretching, flexibility, and cool-down periods, will last for 20 minutes.
  Arms: Standard diaphragm exercise arm

SUMMARY:
This study was designed to investigate and compare the effects of standard diaphragmatic breathing and physiotherapy exercises versus 360-degree expandable diaphragmatic breathing and physiotherapy exercises on respiratory functions, respiratory muscle strength, clinical course of the disease (such as thoracic mobility, flexibility), and functional status in individuals with Ankylosing Spondylitis (AS).

DETAILED DESCRIPTION:
One of the primary problems in Ankylosing Spondylitis (AS) is decreased thoracic expansion. For this reason, breathing exercises, especially thorax expansion, should be included. Moreover, according to Pascal's principle, the pressure applied to a closed fluid must be transmitted to every part of the fluid and to the walls of the space in which it is located, without decreasing (13). For this reason, it is thought that the disrupted breathing pattern cannot be adequately corrected by standard diaphragm exercises, in which the patient's hand is placed on the abdomen and the anterior abdominal wall is pushed forward/outward, and the diaphragm descent to the caudal level during inspiration with 360-degree expansion of the thoraco-abdominal cavity may not be sufficient (14). The aims of this study are as follows:

1. To examine and compare the effects of standard diaphragmatic breathing and physiotherapy exercises and 360-degree expanded diaphragm exercises and physiotherapy exercises on respiratory function in individuals with AS.
2. To examine and compare the effects of standard diaphragmatic breathing and physiotherapy exercises, 360-degree expanded diaphragm exercises and physiotherapy exercises on inspiratory and expiratory muscle strength in individuals with AS.
3. To examine and compare the effects of standard diaphragmatic breathing and physiotherapy exercises, 360-degree expanded diaphragm exercises and physiotherapy exercises on spinal mobility and the clinical course of the disease in individuals with AS.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-60 years
* Diagnosis according to the 1988 Modified New York criteria
* Voluntary participation
* BASDAI score of 3 or 4
* No mental problems that could hinder cooperation and understanding

Exclusion Criteria:

* Presence of a neurological disease
* Other respiratory system diseases that could affect chest expansion (COPD, asthma, etc.)
* Regular exercise within the last 3 months Additionally, individuals who miss four consecutive exercise sessions or require a change in treatment will be excluded from the study.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Spinal movements and spinal mobility | From enrollment to the end of treatment at 6 weeks
  The Bath Ankylosing Spondylitis Metrology Index (BASMI) will be used to measure clinical differences in spinal movements and spinal mobility. BASMI includes five measurements: cervical rotation, tragus-to-wall distance, lateral lumbar flexion, anterior lumbar flexion, and intermalleolar distance. A lower score on the BASMI indicates better spinal mobility (15).

SECONDARY OUTCOMES:
Functional status | From enrollment to the end of treatment at 6 weeks
  The functional status of individuals with ankylosing spondylitis will be assessed using Bath Ankylosing Spondylitis Functional Index (BASFI,0-10 cm).
Respiratory muscle strength | From enrollment to the end of treatment at 6 weeks
  Respiratory muscle strength will be measured using a portable device capable of electronically measuring intraoral pressure (RP Check, MD Diagnostics Ltd., Maidstone, UK). Using the non-invasive method of intraoral pressure measurement, maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) will be recorded.
Expiratory Forced Vital Capacity (FVC) | From enrollment to the end of treatment at 6 weeks
  the maximum amount of air that can forcibly be blown out after full inspiration
Forced Expiratory Volume in one second (FEV1) | From enrollment to the end of treatment at 6 weeks
  FEV1 is the volume of air that can forcibly be blown out in first 1 second after full inspiration.
Forced Expiratory Flow at 25-75% of FVC (FEF25-75%) | From enrollment to the end of treatment at 6 weeks
  Mean of forced expiratory flow over the middle half of the forced vital capacity.
FEV1/FVC ratio (FEV1%) | From enrollment to the end of treatment at 6 weeks
  Ratio of forced expiratory volume in one second to forced vital capacity.
Disease activity | From enrollment to the end of treatment at 6 weeks
  Disease activity will be assessed using Ankylosing Spondylitis Disease Activity Index' in (BASDAI) clinical diagnosis and evaluation of disease activity. This index is used to define the activity, progression, and prognosis of the disease. It is interpreted on a score ranging from 0-10. An increase in the score indicates an increase in disease activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Izmir University of Economics, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No